CLINICAL TRIAL: NCT06749717
Title: Knowledge, Attitude, Behavior and Prevalence of Dental Caries of Rural Mothers and Their Preparatory School Young Adults in El-Sobehy Village, Fayoum, Egypt: a Cross-Sectional Study
Brief Title: Knowledge, Attitude, Behavior and Prevalence of Dental Caries of Rural Mothers and Their Preparatory School Young Adults in El-Sobehy Village, Fayoum, Egypt
Acronym: rural
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Samy Sadek Abdelsamea El Touny, Principal Investigator, Cairo University
Other Study IDs: 14422020449571
Record Dates: First submitted 2024-09-28; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Dental Caries
Keywords: attitude; knowledge; behavior; mothers; young adults; impact; rural mothers; fayoum governorate, egypt; dental caries
MeSH Terms: conditions — Dental Caries; Behavior; Tooth, Impacted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to assess prevalence of dental caries, knowledge, attitude and oral hygiene behavior of mothers and their effect on the oral health knowledge, attitude, behavior and dental caries prevalence of their young adult students in a rural school in El-Sobehy village, at Fayoum Governorate in Egypt.

DETAILED DESCRIPTION:
Introduction:

Scientific background:

Oral health is an essential part of overall health and well-being, with growing data suggesting an association between oral and systemic health for serious disorders including cancer, mild cognitive impairment, arthritis, diabetes and cardiovascular disease. Even though oral health has made enormous strides, the burden of oral health disorders is still quite high globally. This may be primarily due to a lack of healthy oral behaviors that are essential in managing the most prevalent oral diseases, such as dental caries and periodontal disease, with a prevalence rate of up to 47.6% or more in school young adults around the globe.

Dental caries is considered as the major oral problem which affect between 60% and 90% of children, and may reach to 100% of adults. Also, dental caries affect 2.4 billion people around the world. The percentage increases to 35% when all ages are included.

The prevalence of oral diseases continues to increase in most low and middle income countries (LMICs) due to urbanization and changing living conditions, low fluoride exposure and lack of access to basic oral health care. Additionally, poor dietary habits with high sugar content and tobacco consumption also increase the risk of oral diseases.

Preventive knowledge and attitude is the first step to reducing the prevalence of dental caries. Oral hygiene habits play an important role in the development of dental caries, and certain changes can have a significant impact on oral health and the status of caries progress. Patient dental awareness and attitude has been shown to significantly reduce the incidence of dental caries in patients.

The Egyptian Ministry of Health and population, in collaboration with the WHO country office Egypt released results of an epidemiological study on oral health status, which showed that utilization of dental services is not at optimal level. Overall 40% of participants reported that they experienced dental problems at the time of examination but did not see a dentist for treatment. According to participant behavior through the dental visit, over 20% had not seen a dentist in over two years, and another 20% had never gone to one.

Family is the Main Influencer of young adult's environment which affect the development and establishment of oral health behaviors. As a young adult's first instructors, parents are crucial in helping them develop a routine of dental hygiene practices by modeling good health behaviors.

Improvement in young adult's oral health depends on their parents' knowledge, attitude and education level. Parental education is the most commonly-used measures of socioeconomic condition in epidemiological studies on young adult's oral health outcomes.

Parents with more education have a more positive attitude regarding their young adult's oral health and pay more attention to preserving their young adult's healthy dentition. Lower-educated parents have been shown to pay less attention to their young adult's oral care habits and regular dentist visits.

To create and implement an effective young adult's oral health agenda and awareness programs for parents and schoolteachers that will enhance oral health, the prevalence of dental caries should be regularly monitored. Therefore, this study aimed to evaluate the prevalence of dental caries in mothers and their young adults in Fayoum, Egypt, and to evaluate the oral hygiene knowledge in mothers and their young adults by Hiroshima University-Dental Behavioral Inventory (HU-DBI) questionnaire and clinical examination.

Review of literature:

Dental caries is quite common in nations where preventive strategies for oral diseases have not yet been put into place. Few studies about the knowledge, attitude, behavior and prevalence of dental caries among the school students and their mothers in Egypt are available and the determination of the exact burden of dental caries remains a considerable challenge.

In research on the prevalence of dental caries in school young adults, aged 12 to 14 years in Riyadh, it was found that just 6.3% of the entire sample was caries-free, with an estimated 93.7% caries frequency.

one study stated that the stage of tooth affection could determine the followed line of treatment. Moreover, have proved that the ICDAS II system had a higher level of sensitivity for detecting non-cavitated carious lesions in comparison to the DMF index.

Another Study compared the dmft/DMFT and ICDAS indices on young adults/adolescents and their mothers. Their results were consistent with the manifestation of a chronic disease, in young adults and adolescents. There were statistically significant differences because incipient or less severe lesions were more frequent and couldn't be detected by the dmft/DMFT index, which lead to an underestimation of the disease in young adults and losing much information. Moreover; it was of great advantage to use ICDAS system with young adults because it presents a cost-effective method while in adults its use could be analyzed according to the available resources since its cost-effectiveness is lower. For this reason, it is important to consider the use of ICDAS in young adults and adolescents.

Study assessed the knowledge, attitude, and preventive practices of parents in Saudi Arabia in regards to the prevention of ECC. They concluded that parents did not show an adequate knowledge but did show a good attitude and practice regarding the prevention of ECC. It is possible that parents are not properly informed about the details of oral disease and its causes.

Egyptian study evaluated the effect of oral health promotional program on knowledge, attitude and practices regarding dental caries among primary school young adults in Minia city, Egypt. They stated that there was improvement of level of knowledge, positive attitudes and satisfactory practices among the majority of the participants' children after implementation of oral health promotion program.

Further Egyptian study compared and described the prevalence of dental caries among group of Egyptian students. They concluded that the prevalence of dental caries among Egyptian adolescent is high. ICDAS scoring system revealed higher caries prevalence values than DMFS method. ICDAS method is the best choice for the preventive goals, while DMFS is sufficient for clinical purposes.

The last study assessed, among mothers of young adults aged 6-12 years, mothers' knowledge, attitude and dental behavior about their young adult's oral health and evaluated their influence on their young adult's dental caries. They revealed that young adult's oral health is significantly impacted by oral health-related knowledge, attitude and behaviors of their mothers in addition to income and education level.

Matching criteria and allocation ratio:

Each patient participating in the study will be evaluated by (M.S) using one caries assessment index; DMFT.

Variables:

Demographic data:

The participants will be all Egyptians. Both male and female and not married students will be recruited for this study. The mean, standard deviation (SD) values and frequencies of demographic data will be calculated.

Examiners training and calibration:

The oral examination will be performed by six examiners using both scoring systems in an alternating manner; such that each examiner will use one of the two investigated scoring systems for one week to be shifted to the other scoring system in the subsequent week.

Clinical examination:

Students will be examined visually for dental caries by different examiners applying DMFT diagnosis system for each student, so that each student will have examination chart with the two forms. The teeth will be first cleansed using brushes, rubber cups and prophylaxis paste to remove any food remnants and surface stains. Clinical examination will be performed under standardized conditions using plain disposable dental mirrors, WHO probe and the dental unit light.

Dental caries detection methods:

For the DMFT index, the examiners will record a tooth as decayed only if a cavity will have already been evident. A carious surface will be verified once the WHO probe catches upon insertion with moderate and steady pressure, accompanied by presence of soft dentin at the base of the cavity and/or presence of an opacity adjacent to the examined area, indicating an undermined or demineralized enamel .

Questionnaire design:

An Arabic self-administered questionnaire will be used for this study to be completed by mothers. The questionnaire will employ the Hiroshima University-Dental Behavioral Inventory (HU-DBI) questionnaire which will consist of 20 items to evaluate the knowledge, attitudes and behaviors of mothers pertaining to their oral health. A score will be calculated based on the sum of agree/disagree responses by giving one point to each favorable response of good oral health. High scores indicate good oral health attitudes and behaviors.

Addressing potential source of bias:

The risk of bias is minimized starting with the sampling of the patients, all patients who fit the inclusion and exclusion criteria will be included until the specified sample size is reached to minimize selection bias. Following that subgroup analysis will be done after the results are achieved to minimize any chance of randomization bias within the group.

Study size

Statistical methods:

Calculation will be done based on comparing 2 proportions from matched (paired) samples in a prospective study using McNemar test, the α-error level will be fixed at 0.05, and the power will be set at 80%.

The sample size was calculated using StatCalc version 1.4.3 (Epi InfoTM, CDC, Atlanta, Georgia, USA) using the population survey test, implementing 999999 population size, 69.5% prevalence of dental caries in Egypt based on a previous study, 95% of confidence level and 5% margin of error. To be able to represent the preparatory school young adults in EL-Sobehy village at Fayoum Governorate, the calculated sample size was a total of 326 students.

Statistical analysis will be performed using Medcalc software, version 22 for windows (MedCalc Software Ltd, Ostend, Belgium). Continuous data will be presented as mean and standard deviation (SD) or median and range when appropriate. Categorical and binary data will be presented as frequency and percentage. Correlation between risk factors and caries prevalence will be done using Pearson's or Spearman's correlation. The significance level will be set at p ≤ 0.05 and all tests will be two tailed.

ELIGIBILITY:
Inclusion Criteria:

* All students of aged between 12-15 years of target school and their mothers will participate at the current survey and health education program.

Exclusion Criteria:

* All students of aged not between 12-15 years of target school and their mothers will not participate at the current survey and health education program.
* married students

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study design:
  Cross-sectional observational study. 8. Setting: This observational study will be held in the Preparatory School El-Sobehy Village, Fayoum, Egypt.
  B. Participants:
  9a. Eligibility criteria and selection method: All students of aged between 12-15 years of target school and their mothers will participate at the current survey and health education program.
  The participants will be all Egyptians. Both male and female and not married students will be recruited for this study.
Sampling Method: Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of dental caries of mothers and their young adult students | 3 months
  Measures unit (The Decayed, Missing, Filled Tooth Index Permanent teeth). The Decayed, Missing, Filled index score indicates a total caries experience of an individual and it gives equal weight to decayed, missing because of caries, filled tooth, or tooth surface.
  The sum of the number of Decayed, Missing due to caries, and Filled Teeth in the permanent teeth increase, means worst outcome.
  Decayed Teeth (number of Decayed Teeth) Missing Teeth (number of Missing Teeth due to caries) Filled Teeth (number of Filled Teeth)

SECONDARY OUTCOMES:
Knowledge, Attitude and Practice of mothers and their young adult preparatory students | 3 months
  Method of Measurement (with reference): Arabic version of Hiroshima University-Dental Behavioral Inventory (HU-DBI) Questionnaire (Surme and Akman, 2023)
  Unit of Measurement:
  Dichotomous (Agree/Disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Olfat Elsayed main supervisor and outcome assessor, Professor, Study Chair — Conservative Dentistry Department, Faculty of Dentistry, Cairo University
Locations (2):
- Egypt (2):
  - El-Sobehy Village, Fayoum, Egypt, Al Fayyum
  - Elrozzna secondary school, El-Sobehy Village, youssef elsedek, Fayoum governorate, Fayoum Governorate

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bamashmous NO, El Ashiry EA, Alamoudi NM, Qahtan DK, Alamoudi RA, Felemban OM. Oral health related knowledge, attitude and behavior among group of mothers in relation to their primary school children's oral health: a cross-sectional study. J Clin Pediatr Dent. 2024 Jan;48(1):152-162. doi: 10.22514/jocpd.2024.017. Epub 2024 Jan 3. PMID 38239168
- [Background] Tafere Y, Chanie S, Dessie T, Gedamu H. Assessment of prevalence of dental caries and the associated factors among patients attending dental clinic in Debre Tabor general hospital: a hospital-based cross-sectional study. BMC Oral Health. 2018 Jul 4;18(1):119. doi: 10.1186/s12903-018-0581-8. PMID 29973262
- [Background] Poutanen R, Lahti S, Seppa L, Tolvanen M, Hausen H. Oral health-related knowledge, attitudes, behavior, and family characteristics among Finnish schoolchildren with and without active initial caries lesions. Acta Odontol Scand. 2007 Apr;65(2):87-96. doi: 10.1080/00016350601058077. PMID 17453426
- [Background] Petersen PE, Bourgeois D, Ogawa H, Estupinan-Day S, Ndiaye C. The global burden of oral diseases and risks to oral health. Bull World Health Organ. 2005 Sep;83(9):661-9. Epub 2005 Sep 30. PMID 16211157
- [Background] Nethan S, Sinha D, Mehrotra R. Non Communicable Disease Risk Factors and their Trends in India. Asian Pac J Cancer Prev. 2017 Jul 27;18(7):2005-2010. doi: 10.22034/APJCP.2017.18.7.2005. PMID 28749643
- [Background] Murakami K, Kondo N, Ohkubo T, Hashimoto H. The effect of fathers' and mothers' educational level on adult oral health in Japan. Community Dent Oral Epidemiol. 2016 Jun;44(3):283-91. doi: 10.1111/cdoe.12216. Epub 2016 Feb 12. PMID 26871456
- [Background] Mishra A, Pandey RK, Chopra H, Arora V. Oral health awareness in school-going children and its significance to parent's education level. J Indian Soc Pedod Prev Dent. 2018 Apr-Jun;36(2):120-124. doi: 10.4103/JISPPD.JISPPD_1172_17. PMID 29970627
- [Background] Listl S, Galloway J, Mossey PA, Marcenes W. Global Economic Impact of Dental Diseases. J Dent Res. 2015 Oct;94(10):1355-61. doi: 10.1177/0022034515602879. Epub 2015 Aug 28. PMID 26318590
- [Background] Kawamura M, Ikeda-Nakaoka Y, Sasahara H. An assessment of oral self-care level among Japanese dental hygiene students and general nursing students using the Hiroshima University--Dental Behavioural Inventory (HU-DBI): surveys in 1990/1999. Eur J Dent Educ. 2000 May;4(2):82-8. doi: 10.1034/j.1600-0579.2000.040206.x. PMID 11168468
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of untreated caries: a systematic review and metaregression. J Dent Res. 2015 May;94(5):650-8. doi: 10.1177/0022034515573272. Epub 2015 Mar 4. PMID 25740856